CLINICAL TRIAL: NCT06112691
Title: USING ARTIFICIAL INTELLIGENCE FOR MASS SCREENING OF THE DIABETIC RETINOPATHY
Brief Title: ARTIFICIAL INTELLIGENCE FOR MASS SCREENING OF THE DIABETIC RETINOPATHY IN THE CHERNIVTSI REGION (Pilot Study)
Acronym: AIMDR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: Komisarenko Institute of Endocrinology and Metobolism (Other Government); CheckEye LLC (Industry)
Responsible Party: Principal Investigator, Andrii Korol, MD, PhD, MD, PhD, DMedSc, The Filatov Institute of Eye Diseases and Tissue Therapy
Other Study IDs: 24.01.2022
Record Dates: First submitted 2023-10-29; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Fundus photo; Artificail Intelligence; Diabetes Melitus; Screening; CheckEye; Fundus image; nonmydriatic camera
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- main group: diabetes mellitus
  Interventions: Device: taking fundus photos using non-mydriatic fundus camera - FundusScope Rodenstock
- control group: without diagnosis of diabetes mellitus without retinal diseases
  Interventions: Device: taking fundus photos using non-mydriatic fundus camera - FundusScope Rodenstock

INTERVENTIONS:
Device: taking fundus photos using non-mydriatic fundus camera - FundusScope Rodenstock — using artificial intelligence to identify diabetic retinopathy in the early stages using fundus photography.

SUMMARY:
The purpose of this study is to create a patient-centric environment for early detection of DR with AI-driven solutions.

DETAILED DESCRIPTION:
The purpose of this study is to create a patient-centric environment for early detection of DR with AI-driven solutions.

This study is planned as a follow-up. Participants who meet the eligibility criteria will be recruited from sites staffed by the trained photographers. After assessing eligibility and securing written informed consent, fundus photographs will be captured using a nonmydriatic ocular fundus camera. Images will be taken according to a specific RAssbyAI Check Eye's imaging protocol provided to camera operator, and then analyzed by the RAssbyAI Check Eye's. The photography protocol consists of two images of the ocular fundus (one optic disc centered, one fovea centered).

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of Diabetes mellitus as defined by:

   A. Having met the criteria established by either the World Health Organization (WHO) or the American Diabetes Association (ADA) B. Hemoglobin A1c (HbA1c)>= 6.5% based on repeated assessments C. Fasting Plasma Glucose (FPG) >= 126 mg/dL (7.0 mmol/L) based on repeated assessments D. Oral Glucose Tolerance test with 2 hr plasma glucose >= 200 mg/dL (11.1mmol/L) using equivalent of 75g anhydrous glucose dose in water.

   E. Symptoms of hyperglycemia or hyperglycemic crisis with random plasma glucose >=200mg/dL (11.1 mmol/L).
2. Understanding of the Study and willingness and ability to sign informed consent
3. Patient age 18 or above
4. Diagnostic for diabetes: 4a) Type 1 diabetes of a lest 5 years of evolution; or 4b) Type 2 diabetes

   -

Exclusion Criteria:

1. Patients under 18 years of age;
2. Failure to give informed consent;
3. Presence of retinal diseases - acquired disease: age-related macular degeneration (AMD), occlusion of retinal vessels (ORV), etc.; birth defects: coloboma of choroid or optic nerve disc, etc.; hereditary diseases: retinitis pigmentosa, angioid streaks of the retina, etc.
4. A patient who has already undergone treatment (surgery, laser, etc.) for any disease of the retina: age-related macular degeneration (AMD), retinal vascular occlusion (ARV), etc. These patients should be excluded or allocated to a separate group.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 660 participants were planed to include in study, 410 of them had diabetes mellitus and 250 participants were as a control group without diagnosis of diabetes mellitus.
  All participants were selected for the study based on the following inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The accuracy | Baseline-Month 12
  The accuracy of detecting of DR

SECONDARY OUTCOMES:
The percent of invalid images | Baseline-Month 12
  The percent of invalid images for analysing by neural network
The percent of false positive detection of DR | Baseline-Month 12
  The percent of false positive detection of DR in individuals without DR

CONTACTS AND LOCATIONS:
Overall Officials: Andrii MD Korol, PhD, Principal Investigator — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (1):
- The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: No